CLINICAL TRIAL: NCT04649112
Title: A Phase 1 Study of PBCAR19B in Participants With CD19-expressing Malignancies
Brief Title: Dose-escalation Study of Safety of PBCAR19B in Participants With CD19-expressing Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Precision BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBCAR19B-01
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: CD19 Expressing Malignancies; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): In this study, PBCAR19B, allogeneic anti-CD19 CAR T Cells, is used to treat participants with relapsed or refractory (r/r) Non-Hodgkin Lymphoma (NHL).
  Route of Administration: Intravenous injection/infusion.
  Interventions: Genetic: PBCAR19B
- Dose Level 2 (Experimental): In this study, PBCAR19B, allogeneic anti-CD19 CAR T Cells, is used to treat participants with relapsed or refractory (r/r) Non-Hodgkin Lymphoma (NHL).
  Route of Administration: Intravenous injection/infusion.
  Interventions: Genetic: PBCAR19B
- Dose Level 3 (Experimental): In this study, PBCAR19B, allogeneic anti-CD19 CAR T Cells, is used to treat participants with relapsed or refractory (r/r) Non-Hodgkin Lymphoma (NHL).
  Route of Administration: Intravenous injection/infusion.
  Interventions: Genetic: PBCAR19B

INTERVENTIONS:
Genetic: PBCAR19B — Single dose of Allogeneic Anti-CD19 CAR T cells will be injected/infused
  Other Names: Allogeneic Anti-CD19 CAR T cells

SUMMARY:
This is a Phase 1, nonrandomized, open-label, single-dose, dose-escalation, and dose-expansion study to evaluate the safety and clinical activity of PBCAR19B in adult study participants with CD-19 expressing malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD19+ expressing malignancies
* At least 2 prior regimens per Standard of Care

Exclusion Criteria:

* No history of active CNS involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Day 1 - Day 28
  To determine the maximum tolerated dose (MTD)
Number of participants with Dose Limiting Toxicity(ies) | 1 year
  To assess adverse events as dose limiting toxicities as defined by the protocol and CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Vainorius, MD, Study Chair — Precision BioSciences, Inc.
Locations (7):
- United States (7):
  - Banner MDA, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lifespan Cancer Institute at Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No